CLINICAL TRIAL: NCT00996125
Title: Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) 580299 Vaccine in Healthy Chinese Female Subjects
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Human Papillomavirus 580299 Vaccine in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112022
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
Keywords: Immunogenicity; Safety; Human papillomavirus; China; HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of Cervarix vaccine. Cervarix vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: CervarixTM
- Placebo Group (Experimental): Subjects received 3 doses of placebo. Placebo vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Other: Control

INTERVENTIONS:
Biological: CervarixTM — Subjects will receive three doses of the Cervarix vaccine intramuscularly according to a 0, 1, 6-month schedule.
  Arms: Cervarix Group
Other: Control — Subjects will receive three doses of control intramuscularly according to a 0, 1, 6-month schedule.
  Arms: Placebo Group

SUMMARY:
This study is designed to evaluate the immunogenicity and safety of GlaxoSmithKline Biologicals' human papillomavirus (HPV) vaccine in pre-teen and adolescent female subjects aged 9 - 17 years. One group of subjects will receive the HPV vaccine and the other group will receive the control.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they or their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Healthy Chinese females between and including 9 and 17 years of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject and informed assent obtained from the subject, if appropriate, prior to enrolment.
* Healthy subjects as established by medical history and history-directed clinical examination before entering into the study.
* Subjects must not be pregnant. Absence of pregnancy will be verified with a urine pregnancy test before each vaccination.
* Subjects must be either of non-childbearing potential, or if of childbearing potential, they must be abstinent or have practiced adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and agree to continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after (i.e., Days 0-29) the first dose of vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* A subject planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding. Subjects must be at least three months post-pregnancy and not breastfeeding to enter the study.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the protocol during the study period.
* Previous administration of components of the study vaccine.
* History of chronic condition(s) requiring treatment such as cancer or autoimmune disease.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 9 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2009-10-24; Primary Completion 2010-12-08 (Actual); Study Completion 2010-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Zhu F, Li J, Hu Y, Zhang X, Yang X, Zhao H, Wang J, Yang J, Xia G, Dai Q, Tang H, Suryakiran P, Datta SK, Descamps D, Bi D, Struyf F. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine in healthy Chinese girls and women aged 9 to 45 years. Hum Vaccin Immunother. 2014;10(7):1795-806. doi: 10.4161/hv.28702. PMID 25424785
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix Group | Placebo Group
Started | 374 | 376
Completed | 369 | 365
Not Completed | 5 | 11
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 6
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 374 | 376 | 750
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.1 (2.44) | 13.1 (2.42) | 13.1 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 376 | 750
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) for Antibodies Against Human Papillomavirus (HPV)-16/18 Antigens
Description: Titers were given as geometric mean titers and were measured by Enzyme-linked Immunosorbent Assay (ELISA) and expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: One month after the third dose (at Month 7)
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity which included subjects who received 3 doses of the study vaccine or placebo and for whom data concerning immunogenicity measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 362 | 363
EL.U/mL
  Anti-HPV-16 | 18347.1 [16915.2 to 19900.2] | 5.0 [4.7 to 5.3]
  Anti-HPV-18 | 7960.2 [7181.3 to 8823.6] | 4.1 [3.8 to 4.3]

2. Secondary Outcome: Number of Subjects Seroconverted for Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Seroconversion is defined as the appearance of anti-HPV-16 and/or anti- HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the sera of subjects seronegative before vaccination. Cut-off values were 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti- HPV-18 antibodies.
Time Frame: At Month 7
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity on initially seronegative subjects for whom data concerning immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 338 | 344
Participants
  Anti-HPV-16: number analyzed (Participants) | 326 | 323
  Anti-HPV-16 | 326 | 8
  Anti-HPV-18 | 336 | 10

3. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 50 millimeter (mm).
Time Frame: During the 7 days (Days 0 - 6) following each vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 373 | 376
Participants
  Any pain | 350 | 299
  Grade 3 pain | 38 | 16
  Any redness | 113 | 52
  Grade 3 redness | 2 | 1
  Any swelling | 113 | 54
  Grade 3 swelling | 13 | 2

4. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, urticaria and fever (= axillary temperature above 37.0 degrees Celsius (°C). Grade 3 fever = axillary temperature above 39.0°C. Grade 3 urticaria = urticaria distributed on at least 4 body areas. For other symptoms, any = occurrence of any general symptom regardless of intensity grade or relation to vaccination and grade 3 = a general symptom that prevented normal activity. Related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7 days (Days 0 - 6) following each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 373 | 376
Participants
  Any arthralgia | 38 | 33
  Grade 3 arthralgia | 0 | 2
  Related arthralgia | 25 | 23
  Any fatigue | 137 | 126
  Grade 3 fatigue | 2 | 4
  Related fatigue | 106 | 98
  Any gastrointestinal symptoms | 57 | 45
  Grade 3 gastrointestinal symptoms | 2 | 2
  Related gastrointestinal symptoms | 21 | 31
  Any headache | 123 | 99
  Grade 3 headache | 5 | 3
  Related headache | 80 | 70
  Any myalgia | 110 | 93
  Grade 3 myalgia | 1 | 1
  Related myalgia | 96 | 83
  Any rash | 9 | 4
  Grade 3 rash | 0 | 0
  Related rash | 3 | 2
  Any fever | 86 | 74
  Grade 3 fever | 2 | 0
  Related fever | 40 | 27
  Any urticaria | 8 | 3
  Grade 3 urticaria | 0 | 0
  Related urticaria | 7 | 1

5. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions (MSCs)
Description: Medically significant conditions (MSCs) are defined as: adverse events (AEs) prompting emergency room or physician visits that are not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury.
  MSCs were collected regardless of causal relationship to vaccination and intensity.
Time Frame: Throughout the study period (from Day 0 up to Month 12)
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 374 | 376
Participants | 14 | 11

6. Secondary Outcome: Number of Subjects Reporting Pregnancies and Pregnancy Outcomes
Time Frame: Throughout the study period (from Day 0 up to Month 12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 374 | 376
Participants | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: Within 30 days (Days 0 - 29) after any vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 374 | 376
Participants
  Any AEs | 139 | 125
  Grade 3 AEs | 0 | 3
  Related AEs | 2 | 3

8. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Throughout the study period (from Day 0 up to Month 12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 374 | 376
Participants
  Any SAEs | 5 | 2
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Day 0 up to Month 12. Systematically assessed frequent adverse events (AEs) and non-systematically assessed frequent AEs were assessed during 7 days and 30 days post vaccination period respectively.
Description: For the systematically assessed other (non-serious) adverse events, the total participants at risk in Cervarix Group included those from Total Vaccinated cohort who had the symptom sheet completed and with at least one documented dose.
Arm/Group | Cervarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 5/374 | 2/376
Other Adverse Events (participants affected / at risk) | 360/374 | 339/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=374) | Placebo Group (N=376)
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Group (N=374) | Placebo Group (N=376)
Upper respiratory tract infection (Infections and infestations) | 101 | 86
Nasopharyngitis (Infections and infestations) | 22 | 18
Pain (General disorders) | 350/373 | 299
Redness (General disorders) | 113/373 | 52
Swelling (General disorders) | 113/373 | 54
Arthralgia (General disorders) | 38/373 | 33
Fatigue (General disorders) | 137/373 | 126
Gastrointestinal symptoms (General disorders) | 57/373 | 45
Headache (General disorders) | 123/373 | 99
Myalgia (General disorders) | 110/373 | 93
Fever (General disorders) | 86/373 | 74 — Fever is defined as axillary temperate above 37.0 degrees Celsius.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.